CLINICAL TRIAL: NCT06262971
Title: Comprehensive Registry of Left Main Coronary Artery Percutaneous Coronary Intervention Outcomes at Istanbul Medipol University Hospital
Brief Title: Left Main Percutaneous Coronary Intervention Registry in Istanbul Medipol University Hospital
Status: Completed | Type: Observational
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Ozgur Ulas Ozcan, Prof Dr Ozgur Ulas Ozcan, Medipol University
Other Study IDs: PCI-LM-Registry-2018
Record Dates: First submitted 2024-02-08; First posted 2024-02-16 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2024-02

CONDITIONS: Coronary Artery Disease; Left Main Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Percutaneous coronary intervention — balloon angioplasty, stent implantation, atherectomy, intravascular ultrasound.

SUMMARY:
This hospital-based registry study at Istanbul Medipol University Hospital focuses on documenting and analyzing the clinical and demographic characteristics, procedural-related aspects, and both short and long-term outcomes of patients undergoing left main coronary artery percutaneous coronary intervention (PCI). The study aims to identify predictors for adverse clinical outcomes in patients treated for left main coronary artery disease.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing any PCI procedure(s) in given timeframe will be included in this registry

Exclusion Criteria:

* Patients with no informed consent

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients performing any PCI procedure(s) in given timeframe will be included in this registry
Sampling Method: Non-Probability Sample
Enrollment: 3620 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Incidence of Major Adverse Cardiac Events (MACE) within One Year Following Left Main Coronary Artery PCI | up to 1 month, 3 months, 1 year
  The primary outcome measure will be the incidence of major adverse cardiac events (MACE) within one year post-procedure in patients undergoing left main coronary artery PCI. MACE is defined as a composite of clinically significant endpoints including all-cause mortality, non-fatal myocardial infarction, non-fatal stroke, and any revascularization procedures required after the initial PCI.

SECONDARY OUTCOMES:
Ischemia-Driven Target Vessel Revascularization (ID-TVR) Ischemia-Driven Target Vessel Revascularization (ID-TVR) | 1 year
  Revascularization procedure that is performed on a previously treated vessel in patients who have developed ischemia.
Procedure-Related Complications Within 30 Days of PCI | 1 month
  This outcome will document the incidence of procedure-related complications, including bleeding, vascular complications, or acute kidney injury, occurring within 30 days post-PCI.
Health-Related Quality of Life (HRQoL) Scores One Year After PCI | 1 year
  Health-related quality of life using standardized questionnaire (SF-36) one year after the PCI procedure
Rate of stent thrombosis | 1 month, 3 months, 1 year
  Probable or definite stent thrombosis

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medipol University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
Planned after analysis